CLINICAL TRIAL: NCT05382819
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of Single and Multiple Ascending Doses of FRTX-02 in Healthy Subjects and Subjects With Atopic Dermatitis
Brief Title: A Safety, Tolerability and Preliminary Efficacy Study of FRTX-02 Capsules in Healthy Subjects and Subjects With Atopic Dermatitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Fresh Tracks Therapeutics, Inc. (Industry)
Collaborators: Syneos Health (Other); Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BBI-02-101
Record Dates: First submitted 2022-04-04; First posted 2022-05-19 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Atopic Dermatitis Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part 1A Single Ascending Dose (SAD) - Active (Experimental): Increasing dose of FRTX-02 Capsules will be administered to healthy volunteers.
  Interventions: Drug: FRTX-02 Capsule
- Part 1A Single Ascending Dose (SAD) - Placebo (Placebo Comparator): Matching placebo will be administered to healthy volunteers.
  Interventions: Drug: Placebo
- Part 1B Multiple Ascending Dose (MAD) - Active (Experimental): Increasing dose of FRTX-02 Capsules will be administered to healthy volunteers.
  Interventions: Drug: FRTX-02 Capsule
- Part 1B Multiple Ascending Dose (MAD) - Placebo (Placebo Comparator): Matching placebo will be administered to healthy volunteers.
  Interventions: Drug: Placebo
- Part 2 Subjects with Moderate to Severe Atopic Dermatitis (AD) - Active (Experimental): FRTX-02 Capsules will be administered daily for 28 days to subjects with atopic dermatitis.
  Interventions: Drug: FRTX-02 Capsule
- Part 2 Subjects with Moderate to Severe Atopic Dermatitis (AD) - Placebo (Placebo Comparator): Matching placebo will be administered daily for 28 days to healthy volunteers.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FRTX-02 Capsule — DYRK-1A Inhibitor
  Arms: Part 1A Single Ascending Dose (SAD) - Active; Part 1B Multiple Ascending Dose (MAD) - Active; Part 2 Subjects with Moderate to Severe Atopic Dermatitis (AD) - Active
Drug: Placebo — Matching Placebo
  Arms: Part 1A Single Ascending Dose (SAD) - Placebo; Part 1B Multiple Ascending Dose (MAD) - Placebo; Part 2 Subjects with Moderate to Severe Atopic Dermatitis (AD) - Placebo

SUMMARY:
FRTX-02 is an orally-available, potent and selective DYRK1A inhibitor.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, double blind study in healthy subjects and subjects with atopic dermatitis that is designed to assess the safety and tolerability of FRTX-02 capsules at single and multiple ascending doses.

Safety will be assessed through vital signs, ECG, adverse events and safety laboratory tests.

Pharmacokinetic and pharmacodynamic information will also be collected.

ELIGIBILITY:
Selected Inclusion Criteria

Part 1 (SAD/MAD)

* Healthy male or female
* 18-55 years of age, inclusive
* At least 50 kg in weight (males) and 45 kg in weight (females)
* BMI 18.5-30.0 kg/m2, inclusive

Part 2 (Subjects with AD)

* Male or female with atopic dermatitis
* 18-65 years of age, inclusive
* BMI 18-40.0 kg/m2, inclusive
* Validated Investigator's Global Assessment (vIGA-AD) score of ≥ 3 (moderate)
* Body surface area (BSA) with AD involvement ≥ 10%
* History of inadequate response to treatment with topical medications (e.g., corticosteroids, calcineurin inhibitors, etc.) or subjects for whom topical treatments are otherwise medically inadvisable.

Selected Exclusion Criteria

Part 1 (SAD/MAD)

* Use of tobacco products within 3 months prior to drug administration
* History of alcohol abuse or drug abuse
* Positive urine drug screen, alcohol breath test, or urine cotinine test
* Participation in a clinical research study involving the administration of an investigational or marketed drug within 30 days prior to drug administration
* Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to dosing.

Part 2 (Subjects with AD)

* History of alcohol abuse or drug abuse
* Positive urine drug screen, alcohol breath test, or urine cotinine test
* Participation in a clinical research study involving the administration of an investigational or marketed drug within 12 weeks prior to drug administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
The number of participants with treatment-emergent adverse events. | Up to Day 8 (Part A: SAD); up to Day 21 (Part B MAD); up to Day 43 (Part 2)
  Number of participants with adverse events, abnormal vital signs, abnormal ECG readings and abnormal laboratory test results.

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health Quebec, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No